CLINICAL TRIAL: NCT05807776
Title: A Phase II Prospective Study to Evaluate the Safety and Efficacy of Tislelizumab Monotherapy or Combined With Lenvatinib as Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma.
Brief Title: Tislelizumab Monotherapy or Combined With Lenvatinib as Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2211001174
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Resectable Hepatocellular Carcinoma
MeSH Terms: interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tislelizumab (Experimental): Received tislelizumab for 2 cycles, 200mg, iv, d1,Q3W. Patients achieved PR or reduced SD were enrolled in arm 1 and accepted surgery. After surgery, patients in arm 1 would receive tislelizumab as adjuvant therapy for 3-6 months.
  Interventions: Drug: Tislelizumab
- tislelizumab+lenvatinib (Experimental): Received tislelizumab for 2 cycles, 200mg, iv, d1,Q3W. Patients achieved PD or increased SD were enrolled in arm 2 and continued to accept treatment with tislelizumab and lenvatinib for 2 cycles.
  After 2 cycles, patients would receive surgery according to their physical conditions.
  After surgery, patients in arm 2 would receive tislelizumab and lenvatinib as adjuvant therapy for 3-6 months.
  Interventions: Drug: Tislelizumab; Drug: Tislelizumab, Lenvatinib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg, iv, d1, Q3W
Drug: Tislelizumab, Lenvatinib — Tislelizumab combined with lenvatinib:
  Tislelizumab 200mg, iv, d1, Q3W Lenvatinib 8mg，po，qd.
  Arms: tislelizumab+lenvatinib

SUMMARY:
This is a phase II prospective study to evaluate the safety and efficacy of Tislelizumab monotherapy or combined with lenvatinib as neoadjuvant therapy for resectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a known diagnosis of HCC as defined in the protocol
2. Patients must be evaluated by the Department of Hepatobiliary Oncology, Tianjin Medical University Cancer Hospital to determine whether they can complete surgical treatment. Patients can be resectable in both oncology and surgery.
3. At least ≥1 measurable lesion (RECIST 1.1)
4. Age 18-75, male or female
5. ECOG PS 0-1
6. Child-pugh A
7. The function of vital organs meets the following requirements (excluding the use of any blood component and cell growth factor within 14 days)

   Blood routine:

   Neutrophils ≥1.5×109//L Platelet count ≥100×109/L Hemoglobin ≥90g/L

   Liver and kidney function:

   Serum creatinine (SCr) ≤ 1.5 times upper limit of normal value (ULN) or creatinine clearance ≥50 ml/min (Cockcroft-Gault formula) Total bilirubin (TBIL)≤ 1.5 times the upper limit of normal value (ULN) AST or ALT levels ≤ 3 times the upper limit of normal value (ULN)
8. Normal coagulation function, International standardized ratio INR≤1.5×ULN or Prothrombin time PT≤1.5ULN
9. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. Subjects whose baseline TSH is outside the normal range may be enrolled if total T3 (or FT3) and FT4 are within the normal range.
10. Myocardial enzyme profiles were within the normal range (simple laboratory abnormalities that were not clinically significant were also allowed to be included)
11. Patients who have progressed to PD or increased SD after 2 cycles of tislelizumab monotherapy must be willing to continue 2 cycles of tislelizumab and Lenvatinib combination therapy and be evaluated.

Exclusion Criteria:

1. Have received any systemic anticancer therapy or radiotherapy for their current tumor or other primary tumor in the 6 months prior to study entry.
2. Tumor load or tumor growth rate was considered by the investigator to be insufficient to delay surgery.
3. Had major surgery within 14 days prior to neoadjuvant therapy.
4. Uncontrolled co-morbidities defined in the protocol and identified by the investigator.
5. Receiving systemic steroid therapy or any other immunosuppressive therapy within 7 days prior to administration of the first dose of study therapy.
6. Have had an active autoimmune disease requiring systemic treatment within the past 1 year.
7. Have other malignancies that are known, developing and/or require aggressive treatment.
8. Informed consent to encephalitis, meningitis, or uncontrolled seizures in the previous year.
9. A history of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, systemic pneumonia) or active non-infectious pneumonia requires immunosuppressive doses of glucocorticoids to assist in treatment.
10. Bleeding from esophageal or fundus varices caused by portal hypertension in the past 6 months; Severe (G3) varicose veins were known on endoscopy within 3 months prior to initial administration; Patients with evidence of portal hypertension (including imaging findings of a large spleen diameter of more than 10cm and platelets of less than 100) were at high risk of bleeding as assessed by the investigators.
11. History of arteriovenous thromboembolism events within the past 6 months, including myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other severe thromboembolism. Implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis, except in patients with stable thrombus after conventional anticoagulant therapy.
12. Severe bleeding tendency or coagulopathy, or receiving thrombolytic therapy.
13. Prophylactic use of low-dose, low-molecular heparin (e.g., enoxaparin 40 mg/ day) is permitted, except for vitamin K antagonists (e.g., warfarin).
14. Long-term use of drugs that inhibit platelet function such as aspirin, dipyridamole or clopidogrel is required.
15. Uncontrolled hypertension, systolic blood pressure > 140mmHg or diastolic blood pressure > 90 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
16. Symptomatic congestive heart failure (New York Cardiological Association Grade II-IV), symptomatic or poorly controlled arrhythmias, history of congenital long QT syndrome or adjusted QTc > 500ms at screening (calculated using the Fridericia method).
17. A previous history of gastrointestinal perforation and/or fistula within the past 6 months, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive enterectomy (partial resection of the colon or extensive resection of the small intestine with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MPR rate | 4 months
  tumor necrosis rate ≥ 70%

SECONDARY OUTCOMES:
1-year and 2-years DFS% | 36 months
  1-year and 2-years disease-free survival rate
ORR | 3 months
  objective response rate
Surgery delay rate | 3 months
  Surgery was performed more than 28 days after the last cycle of neoadjuvant therapy
MiVI rate | 3 months
  Incidence of microvascular invasion
mOS | 5 years
  Median Overall survival
AE and SAE | 1 year
  adverse reactions

IPD SHARING:
Plan to Share IPD: Yes